CLINICAL TRIAL: NCT06769321
Title: Phase 2 RCT Automatic Thermomechanical Massage Bed for Acute Pain Relief for Chronic Nonspecific Low Back Pain
Brief Title: Automatic Thermomechanical Massage Bed for Acute Pain Relief for Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The City College of New York (Other)
Responsible Party: Principal Investigator, Marom Bikson, Professor, The City College of New York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-0288-CCNY
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: Chronic Pain; Low back Pain; Automatic Thermo-mechanical Therapy
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: This a double-blind sham-controlled randomized trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Automatic Thermomechanical Therapy (Experimental): This device delivers thermomechanical therapy to the lower back for 40 minutes
  Interventions: Device: Automatic Thermo-mechanical Massage Bed
- Sham Automatic Thermomechanical Therapy (Sham Comparator): The comparator device is a sham device that has the same outer appearance as the investigational device. Throughout the entire massage session, the intensity will be set to a level below 1, in areas unrelated to where the major muscles causing lower back pain are located, minimizing the actual massage effect. The thermal component will be turned off entirely.
  Interventions: Device: Automatic Thermo-mechanical Massage Bed

INTERVENTIONS:
Device: Automatic Thermo-mechanical Massage Bed — The MASTER V6 (Master series, CGM MB-1701, CERAGEM Co. Ltd., Cheonan, Korea) used in this study is a commercially available automated thermo-mechanical therapy device that combines mechanical spinal stimulation with far-infrared (FIR) heat treatment.

SUMMARY:
This prospective, double-blinded, sham-control, parallel-arm, randomized pilot trial will recruit n=40 participants, ages 18-65 (inclusive), with chronic low back pain (LBP) in the lower region, to be randomly assigned using 1:1 randomization method to receive a 40-minute single session of either active or sham Automated Thermo-mechanical Therapy (ATT). All research procedures, including informed consent, ATT session, and pre- and post-ATT assessments, will be completed in one single session.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Has had chronic non-specific lower back pain persisting for 12 weeks or more
* Conversational level of English

Exclusion Criteria:

* Contraindications to mechanical manipulation of the back
* History of back surgery within the past three years
* Recent back injury
* Presence of back implants or active implanted devices
* Low back pain resulting from other specific conditions (e.g., infection, neoplasm)
* Sensitivity to heat
* Circulatory insufficiency
* Heart disease
* Pregnant or breastfeeding
* Individuals with a history of substance use disorder
* Body weight over 298 lbs (135 kg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
The 100mm Visual Analogue Scale for Pain | Immediately before and immediately after intervention
  The VAS-P100 is a unidimensional measure of pain intensity, used to record patients' pain progression or compare pain severity between patients. The 100-mm VAS-P is a straight horizontal line of fixed length of 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (best) to the right (worst). The participant marks on the line the point that they feel represents their perception of their current state. The score is determined by measuring in millimeters from the left-hand end of the line to the point that the patient marks

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire | Immediately before intervention
  The Roland-Morris is a 24-item self-report questionnaire about how low-back pain affects functional activities. Total score can range from 0 (no disability) to 24 (severe disability). The RMDQ is scored by adding up the number of items the patient checks.
McGill Pain Questionnaire | Immediately before intervention and immediately after intervention
  This questionnaire is used to evaluate a person experiencing significant pain, to monitor the pain over time and to determine the effectiveness of any intervention. The questionnaire evaluates three different domains: 1) What does the pain look like?; 2) How does your pain change with time?; 3) How strong is your pain?
State-Trait Anxiety Inventory | Immediately before and immediately after intervention
  This questionnaire is widely used to measure the state and trait components of anxiety
5-point Verbal Rating Scale for Pain Relief | Immediately after intervention
  Verbal rating scales about pain relief on a 5-point rating scale: none= 0, slight= 1, moderate= 2, good= 3, complete relief= 4. (Administered only at the post-ATMB intervention)28
Modified-Modified Schöber Test | Immediately before and immediately after intervention
  This is a physical examination used to measure the ability of a patient to flex the lower back. The patient is standing, and the examiner marks both posterior superior iliac spine (PSIS) and then draws a horizontal line at the center of both marks. A second line is marked 15 cm above the first line. The patient is then instructed to flex forward without bending the knees as if attempting to touch his/her toes, examiner re-measures the distance between the top and bottom line

CONTACTS AND LOCATIONS:
Overall Officials: Marom Bikson, PhD, Principal Investigator — The City College of New York
Locations (1):
- The Center for Discovery and Innovation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donnery K, Pilloni G, FallahRad M, Lee K, Han B, Park S, Kim J, Charvet L, Bikson M. Automated thermo-mechanical therapy for immediate relief in chronic non-specific lower back pain: a randomized controlled trial. Front Neuroergon. 2026 Jan 9;6:1674928. doi: 10.3389/fnrgo.2025.1674928. eCollection 2025. PMID 41585325